CLINICAL TRIAL: NCT05821205
Title: Michigan Youth Violence Prevention Center: Building Evidence for Gun Violence Prevention - SafERteens Implementation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patrick Carter, Director, University of Michigan Institute for Firearm Injury Prevention Associate Professor, Department of Emergency Medicine, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00220789; 5-U01-CE-003382-02-00 (Other Grant/Funding Number: Centers for Disease Control and Prevention); 5U01CE003382-02 (NIH)
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-10

CONDITIONS: Violence in Adolescence
Keywords: Gun

STUDY DESIGN:
Intervention Model Description: Providers or staff (n=240) participating in screening (e.g., nurses) and/or intervention delivery (e.g., social workers, child life, community health workers) will be consented/enrolled in the MRT, each person randomized weekly with equal probability to one of three ES or control and also randomized monthly to receive personalized feedback or no personalized feedback.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Narrative Persuasion (randomized weekly, 1 of 4 options) (Experimental): Narrative persuasion will be youth or provider testimonial about violence in their community and/or how SafERteens helped their development and reduced violence. Randomized weekly.
  Interventions: Behavioral: Narrative Persuasion
- Reciprocity (randomized weekly, 1 of 4 options) (Experimental): The reciprocity engagement strategy (ES) will be operationalized as an unsolicited $5 gift card with the SafERteens Logo. Randomized weekly.
  Interventions: Behavioral: Reciprocity
- Commitment (randomized weekly, 1 of 4 options) (Experimental): Commitment will be operationalized as a pledge committing to screening and/or delivering SafERteens (depending on role). Randomized weekly.
  Interventions: Behavioral: Commitment
- Engagement Strategy Control (randomized weekly, 1 of 4 options) (No Intervention): The control condition will involve no ES for the weekly Engagement Strategies. Randomized weekly.
- Personalized feedback control (randomized monthly, 1 of 2 options) (No Intervention): The control condition will involve no personalized feedback. Randomized monthly
- Personalized feedback (randomized monthly, 1 of 2 options) (Experimental): The feedback ES will be operationalized as a visual graphic of their personal performance screening and/or delivering SafERteens in relation to the mean of the provider group and/or towards a pre-set standard (i.e., screening 75% of adolescents; delivery rate of 75% of eligible youth). Personalized feedback or none will be randomized on a monthly basis.
  Interventions: Behavioral: Personalized Feedback

INTERVENTIONS:
Behavioral: Narrative Persuasion — Narratives will use anonymous testimonials from our prior work combined with open-source pictures. The researchers will ask participants to rate the testimonial message as a measure of engagement.
  Arms: Narrative Persuasion (randomized weekly, 1 of 4 options)
Behavioral: Reciprocity — Researchers will track clicking on the gift card as a measure of engagement
  Arms: Reciprocity (randomized weekly, 1 of 4 options)
Behavioral: Personalized Feedback — Researchers will track clicking on a link and/or opening to review visual data as a source of engagement.
  Arms: Personalized feedback (randomized monthly, 1 of 2 options)
Behavioral: Commitment — Providers will receive a commitment message and be asked to reply as a measure of engagement.
  Arms: Commitment (randomized weekly, 1 of 4 options)

SUMMARY:
The purpose of this study is to determine the preliminary efficacy (via a micro-randomized trial [MRT] design) of augmenting Enhanced-Replicating Effective Program (E-REP) with engagement strategies to increase and sustain reach by healthcare providers (e.g., nurses, social workers) during implementation of the SafERteens program across multiple healthcare settings.

DETAILED DESCRIPTION:
This proposal examines whether augmenting the Enhanced-Replicating Effective Program (E-REP) implementation strategy with theory-based engagement strategies (ES) for healthcare providers (i.e., nurses; social workers) improves reach during the implementation of SafERteens across multiple healthcare settings.

SafERteens is a single-session behavioral intervention combining motivational interviewing (MI) and cognitive-behavioral skills training (CBT) shown to reduce multiple violence outcomes, including non-partner (i.e., peer) aggression, non-partner and partner victimization, and violence consequences (e.g., truancy) among emergency department (ED) youth with recent fighting and drinking.

No prior studies have examined the effect of adding individual engagement strategies to an E-REP package or examined the effect of repeatedly applying such strategies over time to enhance implementation of an evidence-based intervention.

In this study, the researchers will test four ES: Narrative Persuasion Strategies, Reciprocity Strategies, Personalized Feedback Strategies, and Commitment Strategies.

The researchers will employ a micro-randomized trial (MRT) design - - a novel experimental design for constructing time-varying m-health interventions. In MRTs, individuals are randomly assigned to intervention options, repeatedly-- at multiple time points over the course of the trial. The data can be used to examine the causal effects of specific ES on a proximal outcome (i.e., reach), changes in these effects over time, and the individual or contextual factors that moderate ES.

In this hybrid type 3 trial, the researchers will embed an MRT testing randomized, weekly delivery of three ES strategies outlined above (and a control option -- no ES) and monthly delivery of Personalized Feedback (and a control option -- No feedback) and will examine preliminary efficacy of those engagement strategies at increasing reach of the implemented SafERteens program. The researchers will also explore potential signals for individual (e.g., age, clinical role), within-individual (e.g., prior engagement), and organizational (e.g., implementation climate) moderators of preliminary ES efficacy, as well as examine comparisons between different ES and trends in their efficacy over time.

This is a portion of a larger study. Although the first consent was signed on February 2023 the clinical trial portion of the study did not start until April 2023. U-M IRBMED initially deemed the study as Exempt from its oversight until September 2023 when U-M IRBMED approved it as a standard study HUM00220789.

ELIGIBILITY:
Inclusion Criteria:

* Employed at study site
* Participate in screening and/or SafERteens delivery.

Exclusion Criteria:

* Would not be expected to complete screening and/or intervention delivery
* Would not begin screening and/or delivering SafERteens within the first 9 months of cohort implementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Preliminary Efficacy: weekly reach by providers | From the start of implementation to 52 weeks or the end of provider's employment if before 52 weeks.
  Reach is defined as the number of participants screened or the number of participants to whom the intervention was delivered.
  The researchers hypothesize that during weeks where providers receive an engagement strategy (ES), reach will be higher than weeks where no ES is received.
Preliminary Efficacy: monthly reach by providers | From the start of implementation to 52 weeks or the end of provider's employment if before 52 weeks.
  Reach is defined as the number of participants screened or the number of participants to whom the intervention was delivered.
  The researchers hypothesize that during months where providers receive personalized feedback, reach will be higher than months where no ES is received.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Carter, MD, Principal Investigator — University of Michigan
Locations (8):
- United States (8):
  - University of Michigan, Ann Arbor, Michigan
  - Trinity Health Medical Group, Academic Family Medicine - Fruitport, Fruitport, Michigan
  - Helen DeVos Children's Hospital Emergency Department, Grand Rapids, Michigan
  - Muskegon Pediatrics, Muskegon, Michigan
  - HealthWest Youth and Family Services, Muskegon, Michigan
  - Hackley Community Care Medical Services, Muskegon, Michigan
  - Trinity Health - Community Health And Well-Being, Muskegon, Michigan
  - Trinity Health-Emergency Department, Muskegon, Michigan

IPD SHARING:
Plan to Share IPD: No